CLINICAL TRIAL: NCT06380491
Title: Impact of Melatonin Treatment on Blood Pressure Circadian Rhythm, Sleep and Metabolic Variables.
Brief Title: Melatonin's Effect on Nighttime Blood Pressure and Sleep in OSA Patients (MEBP-OSA)
Acronym: MEBP-OSA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); Emory University (Other)
Responsible Party: Principal Investigator, Matilde Valencia-Flores, Coordinator/ Head of the Sleep Disorders Clinic, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REF.2338; UNAM-PAPIIT 32-IN216919 (Other: Universidad Nacional Autonoma de Mexico (UNAM))
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Circadian Blood Pressure Rhythm; Obstructive sleep apnea; Melatonin
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Melatonin; Tablets

STUDY DESIGN:
Intervention Model Description: Patients with a non-dipper pattern in blood pressure will randomly enter one of two options: 1) usual medical treatment; 2) treatment with melatonin plus usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care for nocturnal non-dipping Blood Pressurem in OSA (Experimental): 1. Group of participants receives an intervention/treatment considered to be usual care
  Interventions: Drug: Melatonin 3 MG Oral Tablet
- Oral administration of 3 mg/day of melatonin for 30 days in non-dipping Blood Pressure in OSA (Experimental): 2. Group of participants receives oral Melatonin 3 mg/day during 30 days plus usual care
  Interventions: Drug: Melatonin 3 MG Oral Tablet

INTERVENTIONS:
Drug: Melatonin 3 MG Oral Tablet — Participants with OSA and nocturnal non-dipping Blood Pressure will be randomly assigned to a treatment with melatonin 3mg/d or to receive only the usual care.
  Other Names: Usual Care for participants with OSA and nocturnal non-dipping Blood Pressure

SUMMARY:
The goal of this clinical trial is to learn if melatonin works to treat comorbid insomnia in adults with OSA and nocturnal non-dipping blood pressure pattern.

The main question it aims to answer is:

Does melatonin maintain sleep during night and recover the dipping blood pressure pattern?

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if melatonin works to treat comorbid insomnia in adults with OSA and nocturnal non-dipping blood pressure pattern.

The main question it aims to answer is:

Does melatonin maintain sleep during night and recover the dipping blood pressure pattern?

Participants will:

* Take melatonin or the habitual treatment every day for one month
* Visit the clinic 11 times for one month
* Keep a diary of their symptom and activities and use twice a 24 h ambulatory blood pressure monitoring (ABPM), attend two overnight polysomnography studies, and use an actigraph every day for 2 weeks.

Researchers will compare melatonin to the habitual treatment to see if melatonin works to treat insomnia and recover the dipping blood pressure pattern.

The medical problems that participants would have when taking melatonin are:

* changes in blood pressure and cholesterol
* Increased risk of contracting immune system disorders
* Possible increased risk of liver damage.

ELIGIBILITY:
Inclusion Criteria:

* Polisomnographic diagnosis of Obstructive Sleep Apnea
* Non-dipping blood pressure on Ambulatory blood pressure monitoring (ABPM):

Exclusion Criteria:

* Use of sleep or psychiatric medication
* Use of Positive Airway Pressure (CPAP or Bipap)
* Neurologic or psychiatric disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2025-01-22 (Estimated)

PRIMARY OUTCOMES:
Melatonin at a dose of 3 mg before sleep time, after a period of 30 days changes the time awake after sleep onset (WASO), and recovers the dipper pattern of blood pressure | 30 days
  Wake after sleep onset (WASO) and non-dipper patter of Blood Pressure change after melatonin intake for 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Matilde Valencia-Flores, PhD, Principal Investigator — National Institute of Medical Sciences and Nutrition Salvador Zubirán (INCMNSZ)
Locations (1):
- National Institute of Medical Sciences and Nutrition Salvador Zubirán (INCMNSZ), Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Influence of circadian time of hypertension treatment on cardiovascular risk: results of the MAPEC study. Chronobiol Int. 2010 Sep;27(8):1629-51. doi: 10.3109/07420528.2010.510230. PMID 20854139
- [Result] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Blunted sleep-time relative blood pressure decline increases cardiovascular risk independent of blood pressure level--the "normotensive non-dipper" paradox. Chronobiol Int. 2013 Mar;30(1-2):87-98. doi: 10.3109/07420528.2012.701127. Epub 2012 Oct 5. PMID 23039824
- [Result] O'Brien E, Sheridan J, O'Malley K. Dippers and non-dippers. Lancet. 1988 Aug 13;2(8607):397. doi: 10.1016/s0140-6736(88)92867-x. No abstract available. PMID 2899801
- [Result] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Result] Boggia J, Li Y, Thijs L, Hansen TW, Kikuya M, Bjorklund-Bodegard K, Richart T, Ohkubo T, Kuznetsova T, Torp-Pedersen C, Lind L, Ibsen H, Imai Y, Wang J, Sandoya E, O'Brien E, Staessen JA; International Database on Ambulatory blood pressure monitoring in relation to Cardiovascular Outcomes (IDACO) investigators. Prognostic accuracy of day versus night ambulatory blood pressure: a cohort study. Lancet. 2007 Oct 6;370(9594):1219-29. doi: 10.1016/S0140-6736(07)61538-4. PMID 17920917
- [Result] Hansen TW, Li Y, Boggia J, Thijs L, Richart T, Staessen JA. Predictive role of the nighttime blood pressure. Hypertension. 2011 Jan;57(1):3-10. doi: 10.1161/HYPERTENSIONAHA.109.133900. Epub 2010 Nov 15. PMID 21079049
- [Result] Kario K, Kanegae H, Tomitani N, Okawara Y, Fujiwara T, Yano Y, Hoshide S. Nighttime Blood Pressure Measured by Home Blood Pressure Monitoring as an Independent Predictor of Cardiovascular Events in General Practice. Hypertension. 2019 Jun;73(6):1240-1248. doi: 10.1161/HYPERTENSIONAHA.118.12740. PMID 31006331
- [Result] de la Sierra A, Redon J, Banegas JR, Segura J, Parati G, Gorostidi M, de la Cruz JJ, Sobrino J, Llisterri JL, Alonso J, Vinyoles E, Pallares V, Sarria A, Aranda P, Ruilope LM; Spanish Society of Hypertension Ambulatory Blood Pressure Monitoring Registry Investigators. Prevalence and factors associated with circadian blood pressure patterns in hypertensive patients. Hypertension. 2009 Mar;53(3):466-72. doi: 10.1161/HYPERTENSIONAHA.108.124008. Epub 2009 Jan 26. PMID 19171788
- [Result] Eguchi K, Pickering TG, Hoshide S, Ishikawa J, Ishikawa S, Schwartz JE, Shimada K, Kario K. Ambulatory blood pressure is a better marker than clinic blood pressure in predicting cardiovascular events in patients with/without type 2 diabetes. Am J Hypertens. 2008 Apr;21(4):443-50. doi: 10.1038/ajh.2008.4. Epub 2008 Feb 21. PMID 18292756
- [Result] Fagard RH, Thijs L, Staessen JA, Clement DL, De Buyzere ML, De Bacquer DA. Night-day blood pressure ratio and dipping pattern as predictors of death and cardiovascular events in hypertension. J Hum Hypertens. 2009 Oct;23(10):645-53. doi: 10.1038/jhh.2009.9. Epub 2009 Feb 19. PMID 19225527
- [Result] Afsar B, Sezer S, Elsurer R, Ozdemir FN. Is HOMA index a predictor of nocturnal nondipping in hypertensives with newly diagnosed type 2 diabetes mellitus? Blood Press Monit. 2007 Jun;12(3):133-9. doi: 10.1097/MBP.0b013e3280b08379. PMID 17496462
- [Result] Loredo JS, Ancoli-Israel S, Dimsdale JE. Sleep quality and blood pressure dipping in obstructive sleep apnea. Am J Hypertens. 2001 Sep;14(9 Pt 1):887-92. doi: 10.1016/s0895-7061(01)02143-4. PMID 11587154
- [Result] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S13-S28. doi: 10.2337/dc19-S002. PMID 30559228
- [Result] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement D, Coca A, De Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen S, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder R, Shlyakhto E, Tsioufis K, Aboyans V, Desormais I; List of authors/Task Force members:. 2018 Practice Guidelines for the management of arterial hypertension of the European Society of Hypertension and the European Society of Cardiology: ESH/ESC Task Force for the Management of Arterial Hypertension. J Hypertens. 2018 Dec;36(12):2284-2309. doi: 10.1097/HJH.0000000000001961. No abstract available. PMID 30379783
- [Result] Gijon-Conde T, Gorostidi M, Banegas JR, de la Sierra A, Segura J, Vinyoles E, Divison-Garrote JA, Ruilope LM. [Position statement on ambulatory blood pressure monitoring (ABPM) by the Spanish Society of Hypertension (2019)]. Hipertens Riesgo Vasc. 2019 Oct-Dec;36(4):199-212. doi: 10.1016/j.hipert.2019.05.002. Epub 2019 Jun 6. Spanish. PMID 31178410
- [Result] Bastos JM, Bertoquini S, Polonia J. Prognostic significance of ambulatory arterial stiffness index in hypertensives followed for 8.2 years: its relation with new events and cardiovascular risk estimation. Rev Port Cardiol. 2010 Sep;29(9):1287-303. English, Portuguese. PMID 21179973
- [Result] Vaile JC, Stallard TJ, al-Ani M, Jordan PJ, Townend JN, Littler WA. Sleep and blood pressure: spontaneous baroreflex sensitivity in dippers and non-dippers. J Hypertens. 1996 Dec;14(12):1427-32. doi: 10.1097/00004872-199612000-00007. PMID 8986925
- [Result] Aung AT, Chan SP, Kyaing TT, Lee CH. Diabetes mellitus is associated with high sleep-time systolic blood pressure and non-dipping pattern. Postgrad Med. 2020 May;132(4):346-351. doi: 10.1080/00325481.2020.1745537. Epub 2020 Mar 24. PMID 32208051
- [Result] Nikolaidou B, Anyfanti P, Gavriilaki E, Lazaridis A, Triantafyllou A, Zarifis H, Mastrogiannis K, Tsapas A, Douma S, Gkaliagkousi E. Non-dipping pattern in early-stage diabetes: association with glycemic profile and hemodynamic parameters. J Hum Hypertens. 2022 Sep;36(9):805-810. doi: 10.1038/s41371-021-00587-4. Epub 2021 Aug 16. PMID 34400769
- [Result] Pio-Abreu A, Moreno H Jr, Drager LF. Obstructive sleep apnea and ambulatory blood pressure monitoring: current evidence and research gaps. J Hum Hypertens. 2021 Apr;35(4):315-324. doi: 10.1038/s41371-020-00470-8. Epub 2021 Jan 7. PMID 33414503
- [Result] Cuspidi C, Tadic M, Sala C, Gherbesi E, Grassi G, Mancia G. Blood Pressure Non-Dipping and Obstructive Sleep Apnea Syndrome: A Meta-Analysis. J Clin Med. 2019 Sep 2;8(9):1367. doi: 10.3390/jcm8091367. PMID 31480717
- [Result] Pinilla L, Benitez ID, Gracia-Lavedan E, Torres G, Minguez O, Aguila M, Targa A, Dalmases M, Mediano O, Masa JF, Masdeu MJ, Barbe F, Sanchez-de-la-Torre M. Polysomnographic characterization of circadian blood pressure patterns in patients with obstructive sleep apnea. Sleep. 2023 Apr 12;46(4):zsad031. doi: 10.1093/sleep/zsad031. PMID 36806948